CLINICAL TRIAL: NCT06454435
Title: Sintilimab Combined With Fruquintinib and Chemotherapy Versus Sintilimab and Chemotherapy for Conversion Therapy in Unresectable Stage IV Gastric Cancer: a National Multicenter Randomized Controlled Study
Brief Title: Conversion Therapy of Sintilimab in Combination With Fruquintinib and Chemotherapy Versus Sintilimab and Chemotherpay in Stage IV Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20231573
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; S 1 (combination); 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab + Fruquinitinib + S-1 plus nab-paclitaxel (Experimental)
  Interventions: Drug: Sintilimab + Fruquinitinib + S-1 plus nab-paclitaxel
- Sintilimab + S-1 plus nab-paclitaxel (Active Comparator)
  Interventions: Drug: Sintilimab + S-1 plus nab-paclitaxel

INTERVENTIONS:
Drug: Sintilimab + Fruquinitinib + S-1 plus nab-paclitaxel — Drug: Sintilimab Sintilimab 200mg, D1, IV, Q3W 4-8 cycles Drug: Fruquintinib Fruquinitinib 4mg/d, QD, PO, D1-D14, Q3W 4-8 cycles Drug: S-1 BSA<1.25 m2, 40mg twice/day; BSA 1.25-1.5m2, 50mg twice/day; BSA≥1.5 m2, 60mg twice/day, po, D1-D14, Q3W 4-8 cycles Drug: Nab-paclitaxel
  * without peritoneal metastases: 260 mg/m2, IV, D1 for 3h, Q3W 4-8 cycles;
  * with peritoneal metastases: 80mg/m2 IP, plus 180mg/m2, IV, D1, Q3W 4-8 cycles.
  Arms: Sintilimab + Fruquinitinib + S-1 plus nab-paclitaxel
Drug: Sintilimab + S-1 plus nab-paclitaxel — Drug: Sintilimab Sintilimab 200mg, D1, IV, Q3W 4-8 cycles Drug: S-1 BSA<1.25 m2, 40mg twice/day; BSA 1.25-1.5m2, 50mg twice/day; BSA≥1.5 m2, 60mg twice/day, po, D1-D14, Q3W 4-8 cycles Drug: Nab-paclitaxel
  * without peritoneal metastases: 260 mg/m2, IV, D1 for 3h, Q3W 4-8 cycles;
  * with peritoneal metastases: 80mg/m2 IP, plus 180mg/m2, IV, D1, Q3W 4-8 cycles.
  Arms: Sintilimab + S-1 plus nab-paclitaxel

SUMMARY:
This is a multicenter, randomized, open-label, phase 2 clinical study aiming to evaluate the feasibility and efficacy of sintilimab (PD-1 inhibitor) in combination of fruquintinib and chemotherapy (S-1 plus nab-paclitaxel) versus sintilimab and chemotherapy as conversion therapy in patients with stage IV gastric cancer in China.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric/gastroesophageal junction adenocarcinoma through gastroscopy.
* Ages: 18-70 Years (concluding 18 and 70 Years)
* Life expectancy ≥3 months.
* Treatment-naive Stage IV (clinical staging, AJCC 8th) unresectable patients, no prior antitumor therapy (including radiation, chemotherapy, targeted therapy or immunotherapy, etc.).
* The Eastern Cooperative Oncology Group Performance status (ECOG PS) of 0-1.
* Preoperative examinations using CT, MRI, PET-CT, etc., indicating only one unresectable factor OR peritoneal metastasis with another unresectable factor, such as:

  1. N3 lymph node metastasis, mainly referring to group 16 lymph node metastasis.
  2. Extensive or bulky lymph nodes (D2)
  3. Locally advanced T4b.
  4. Hepatic metastases (H1): ≤5 lesions with a total diameter ≤8cm.
  5. Peritoneal metastasis (CY1, P1).
  6. Ovarian metastasis (Krukenberg tumor).
* Physically fit for major abdominal surgery.
* Adequate organ and marrow function, defined as:

  1. Hematological status: Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥100×10^9/L; Hemoglobin (HGB) ≥9.0 g/dL.
  2. Liver function: For patients without liver metastasis, serum total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); ALT and AST ≤2.5×ULN. For patients with liver metastasis: TBIL ≤1.5×ULN; ALT and AST ≤5×ULN.
  3. Renal function: Creatinine clearance (Ccr) ≥50 mL/min (calculated using the Cockcroft/Gault formula).
* Adequate coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 times ULN.
* Voluntary participation and signed informed consent with expected good compliance and follow-up.
* Not involved in other clinical trials.
* Willing to provide blood and histological samples.
* No serious conditions affecting anesthesia, or surgery.
* No hematologic disorders affecting postoperative hemoglobin levels.

Exclusion Criteria:

* Has distal metastases other than oligometastases as defined in the inclusion criteria, such as pulmonary metastases, brain metastases, bone metastases, etc.
* HER-2 positive patients or willing to receive Trastuzumab.
* Endoscopic signs of active bleeding from the lesion.
* Patients with moderate/large volume of ascites.
* Near-obstruction at the cardia or pylorus affecting feeding and gastric emptying or difficulty swallowing tablets.
* Concurrently suffering from other serious illnesses that are difficult to control (Severe uncontrolled recurrent infections, atrial fibrillation, angina pectoris, cardiac insufficiency, ejection fraction measurement under 50%, uncontrolled hypertension, renal insufficiency, symptomatic peripheral neuropathy, and NCI classification >II)
* Has already on other medications prior to enrollment or could not be assured of compliance after enrollment.
* Allergy to any drugs in the regimen.
* Women who are pregnant or breastfeeding and have childbearing potential but are not taking adequate contraceptive measures.
* Organ transplant recipients requiring immunosuppression.
* Patients without decision-making capacity or with psychiatric disorders.
* Systemic treatment with Chinese herbal anti-tumor or immunomodulatory drugs (including thymosin, interferons, interleukins) within 2 weeks before the first dose.
* Use of immunosuppressive drugs within 4 weeks before the first study treatment, excluding local steroids or physiological doses of systemic steroids.
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study treatment.
* Has a diagnosis of autoimmune disease within the previous 2 years (Patients with vitiligo, psoriasis, alopecia areata, or Graves' disease who do not require systemic therapy within the last 2 years, hypothyroidism requiring only thyroid hormone replacement therapy, and type I diabetes mellitus requiring only insulin replacement therapy are eligible for enrollment).
* Known history of primary immunodeficiency.
* Known to have active tuberculosis.
* Has history of human immunodeficiency virus (HIV) infection (i.e., HIV antibody . positive); untreated acute or chronic active hepatitis B or hepatitis C infection. Patients receiving antiretroviral therapy are eligible for enrollment on an individual basis as determined by the physician with monitoring of viral copy number.
* Urinalysis indicating urine protein ≥2+ and 24-hour urine protein quantification >1.0g.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
R0-surgery conversion rate | about 3 years
  The proportion of patients who underwent R0 surgery among all efficacy evaluable patients.

SECONDARY OUTCOMES:
Pathological complete response (pCR) | about 3 years
  The proportion of patients with a pathological complete response (ypT0&N0) at the time of definitive surgery among all patients who underwent conversation surgery.
Major pathological response rate (MPR) | about 3 years
  The proportion of patients with a major pathological response (≤10% residual viable tumor) at the time of definitive surgery among all patients who underwent conversation surgery.
Rate of downstaging | about 3 years
  To determine the rate of ypT0 and ypN0, and downstaging ratio of preoperative imaging clinical stage compared with baseline.
Objective response rate (ORR) | about 3 years
  The proportion of patients who achieved complete response (CR) or partial response(PR) per RECIST v1.1.
Disease control rate (DCR) | about 3 years
  The proportion of patients who achieved CR, PR or stable disease(SD) per RECIST v1.1.
Overall survival (OS) | about 3 years
  The time from the initial date of conversation therapy to the date of death due to any cause.
Progression-free survival (PFS) | about 3 years
  The time from the initial date of conversation therapy to the date of first documentation of disease progression or death due to any cause, whichever occurs first.
Adverse event (AEs) | about 3 years
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Incidence and grade of surgery-related complications will also be as assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China